CLINICAL TRIAL: NCT06007157
Title: Effects of Sodium Glucose Cotransporter-2 Inhibitors on Salt-sensitivity in Patients With Type 2 Diabetes
Brief Title: Sodium Glucose Cotransporter-2 Inhibitors and Salt-sensitivity in Type 2 Diabetes
Acronym: SALT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Andrea Natali, Full Professor of Nutrition, Azienda Ospedaliero, Universitaria Pisana
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SALT
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Blood Pressure; Salt; Excess; Diabete Type 2
Keywords: Salt sensitivity; Sodium glucose cotransporter 2 inhibitors; Type 2 Diabetes; Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2i-treated patients (Experimental)
  Interventions: Behavioral: Hypersodic/Hyposodic diet
- Non SGLT2i-treated patients (Active Comparator)
  Interventions: Behavioral: Hypersodic/Hyposodic diet

INTERVENTIONS:
Behavioral: Hypersodic/Hyposodic diet — Participants will undergo a dietary intervention consisting of a week of high-sodium diet (4800 mg/day), followed by a week of low-sodium diet (1200 mg/day).

SUMMARY:
The goal of this interventional study is to test whether sodium-glucose cotransporter 2 inhibitors (SGLT2i) reduce the effects of high dietary sodium intake in patients with type 2 diabetes.

Participants will undergo a dietary intervention consisting of a week of high-sodium diet, followed by a week of low-sodium diet. At the end of each week the patients will undergo:

* 24-h ambulatory blood pressure measurement;
* 24-h urine collection;
* bioimpedance analysis for body composition determination;
* blood and urine tests.

The study will compare patients treated with SGLT2i and patients not treated with SGLT2i to test whether the treatment reduces the effects of high sodium intake on blood pressure, body composition and biochemical variables.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years;
* both males and females;
* type 2 diabetes.

Exclusion Criteria:

* type 1 diabetes;
* insulin treatment;
* uncontrolled hypertension (SBP > 160 mmHg and/or DBP >95 mmHg);
* pregnancy;
* other acute or chronic conditions influencing blood pressure and glucose metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
24-hour Blood Pressure | 2 weeks
  Systolic and diastolic blood pressure will be measured by 24-h ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Sodium excretion | 2 weeks
  24-hour sodium excretion will be measured by urine collection
Hydration state | 2 weeks
  Hydration state with extra- and intracellular water estimation will be measured by bioimpedance

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with other researchers only upon reasonable request to the PI